CLINICAL TRIAL: NCT02175563
Title: Tilt Cardiopulmonary Resuscitation With a Feedback Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Jaehoon Oh, Department of Emergency Medicine, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Tilt CPR
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Cardiopulmonary Resuscitation; Basic Cardiac Life Support
Keywords: Chest; Compression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Without feedback (No Intervention): Participants compress the chest of the manikin without smartphone based feedback app.
- With feedback (Experimental): Participants compress the chest of the manikin with a smartphone based feedback app.
  Interventions: Device: Audiovisual feedback from smartphone based app

INTERVENTIONS:
Device: Audiovisual feedback from smartphone based app
  Arms: With feedback

SUMMARY:
According to the European Resuscitation Council (ERC) Guidelines for patient to a depth of approximately 5-6 cm on a firm and flat surface when possible. However, Cardiopulmonary resuscitation (CPR) performers may need to continue the chest Resuscitation 2010, CPR performers should compress the sternum of a compression in an oblique direction, such as in elevators. For a pregnant patient in cardiac arrest, the 2010 ERC Guidelines recommend that the performer place the patient in a left-lateral tilt of 15 - 30° using a firm wedge to support the pelvis and thorax because the pregnant uterus can compress the inferior vena cava. We hypothesized Smartphone based chest compression feedback app would improves quality of CPR in an angulated surface.

ELIGIBILITY:
Inclusion Criteria:

* Healthy person
* > 18 years old
* Basic life support educated person

Exclusion Criteria:

* Cardiovascular disease
* Musculoskeletal disease
* Psychiatric disease
* Pregnant
* > 65 years old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Chest compression depth | within the first 30 days after the end of recording
  To measure chest compression depth during 2 minutes
Chest compression rate | within the first 30 days after the end of recording
  To measure the chest compression rate during 2 minutes

SECONDARY OUTCOMES:
Accurate chest compression | within the first 30 days after the end of recording
  To measure the percentage of accurate chest compressions (i.e. correct depth, hand position, and recoil) of total chest compressions during 2 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University, College of medicine, Seoul, South Korea